CLINICAL TRIAL: NCT02563977
Title: Structural Changes In The Abdominal Wall After Deep Inferior Epigastric Perforator Flap Breast Reconstruction
Brief Title: Changes To The Abdominal Wall After DIEP Flap Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kim Alexander Tønseth, Head of Department, Oslo University Hospital
Other Study IDs: KATønseth
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Breast Reconstruction; Abdominal Wall Morbidity
Keywords: Breast reconstruction; Deep inferior epigastric perforator flap; Abdominal wall morbidity; Plastic and reconstructive surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- DIEP flap breast reconstruction: 14 patients who have had DIEP flap breast reconstruction and preoperative CT scan of the abdomen
  Interventions: Device: 2 year postop CT scan of the abdomen

INTERVENTIONS:
Device: 2 year postop CT scan of the abdomen — CT scan of the abdomen (from the xiphoid process to the symphysis) performed approximately two years after performed DIEP flap breast reconstruction. No contrast used. Low dose of radiation.

SUMMARY:
The purpose of this study was to perform an evaluation of the structural changes in the abdominal wall after harvesting a DIEP flap in breast reconstruction.

14 women undergoing secondary, unilateral breast reconstruction were recruited to the study and underwent a 2 year postoperative CT scan of the abdomen (without contrast).

Structural changes were assessed by comparing the abdominal CT scans performed prior to surgery with the 2 year postoperative CT scans.

DETAILED DESCRIPTION:
The purpose of this study was to perform an evaluation of the structural changes in the abdominal wall after harvesting a DIEP flap in breast reconstruction.

14 women undergoing secondary, unilateral breast reconstruction were recruited to the study and underwent a 2 year postoperative CT scan of the abdomen (without contrast).

Structural changes were assessed by comparing the abdominal CT scans performed prior to surgery with the 2 year postoperative CT scans.

The following structural changes were evaluated at four specific levels of the abdomen by two radiologists (among the authors): 1) rectus diastasis, 2) thickness and width of the rectus muscles, 3) thickness of the adipose tissue, 4) hernias (in the zone between the xiphoid process and the symphysis).

The measurement levels chosen were: 1) 7 cm below the xiphoid process, 2) umbilicus level, 3) "central zone" (between level 2 and 4), 4) 5 cm above the symphysis

Statistical analysis were performed to see if the structural measurements were significantly different comparing preoperative CT versus 2 year postoperative CT.

ELIGIBILITY:
Inclusion Criteria:

* Secondary, unilateral breast reconstruction with a DIEP flap
* All smokers stopped smoking 4 weeks prior to surgery

Exclusion Criteria:

* Metastatic disease
* Bilateral breast reconstruction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 14 women consecutively undergoing secondary, unilateral breast reconstruction with a DIEP flap were identified and recruited to participate in the study. The patients were informed about of risks and benefits and gave written consent prior to participation. All smokers stopped smoking 4 weeks prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Structural measurements of the abdominal wall evaluated on CT scans | 2 year postoperative after performed DIEP flap breast reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Tønseth, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Department of Plastic and Reconstructive Surgery, Oslo, Norway